CLINICAL TRIAL: NCT05755828
Title: Prospective, Multicenter, Open, One-arm Clinical Study of Safety and Efficacy of Autologous Stem Cell Transplantation + Anti-CD19 CAR T Cells for B-cell Lymphoma
Brief Title: Clinical Study of Autologous Stem Cell Transplantation + Anti-CD19 CAR T Cells for B-cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2022-KL480-02
Record Dates: First submitted 2023-02-23; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: B-cell Lymphoma
Keywords: Anti-CD19 CAR-T; Autologous stem cell transplantation; Combination therapy
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ASCT+CAR-T Cell Infusion (Experimental): CD19 CAR-T cells were prepared from peripheral lymphocytes of NHL patients with PR after 3 to 4 courses of chemotherapy, and autologous stem cells were collected and frozen after mobilization of patient stem cells by granulocyte stimulating factor (10μg/kg/d*5d). BEAM pretreatment was performed. Autologous stem cells were injected 24 h after pretreatment, and the number of CD34+ cells was > 2*106/kg. On the 6th day after transplantation, autologous Anti-CD19 CAR T cells were transfused, and the dose was determined by the investigator according to the subjects' own disease conditions and in vitro preparation. The patients were given constant intravenous drip/push infusion for 30 minutes.
  Interventions: Biological: ASCT+CAR-T Cell Infusion

INTERVENTIONS:
Biological: ASCT+CAR-T Cell Infusion — CD19 CAR-T cells were prepared from peripheral lymphocytes of NHL patients with PR after 3 to 4 courses of chemotherapy, and autologous stem cells were collected and frozen after mobilization of patient stem cells by granulocyte stimulating factor (10μg/kg/d*5d). BEAM pretreatment was performed. Autologous stem cells were injected 24 h after pretreatment, and the number of CD34+ cells was > 2*106/kg. On the 6th day after transplantation, autologous Anti-CD19 CAR T cells were transfused, and the dose was determined by the investigator according to the subjects' own disease conditions and in vitro preparation. The patients were given constant intravenous drip/push infusion for 30 minutes.

SUMMARY:
To evaluate the CR rate of B-NHL subjects who achieved PR at intermediate assessment after first-line chemotherapy treated with autologous stem cell transplantation + Anti-CD19 CAR T cells.

DETAILED DESCRIPTION:
At present, the incidence of malignant hematological diseases represented by leukemia, lymphoma and multiple myeloma is increasing year by year, ranking in the top ten of tumor incidence and mortality, which greatly endangers people's health and social development . B-cell non-Hodgkin's lymphoma (NHL) is a common aggressive malignant lymphoma. Poor response of some patients to traditional first-line chemotherapy is one of the major problems facing this disease. As a result, researchers are using emerging tools such as high-throughput sequencing to further understand the nature of the disease, refine the classification of the disease, and on this basis develop personalized treatments to improve the prognosis of the disease.

Lymphoma has a complex immunosuppressive microenvironment that may prevent CAR T from achieving sustained precision tumor killing. As a revolutionary immunotherapy strategy, CAR-T therapy is currently faced with some bottleneck problems such as post-treatment relapse (including antigen loss relapse and antigen positive relapse), CAR-T consumption, off-target effect and so on.

At present, autologous stem cell transplantation still plays a pivotal role in high-risk B-NHL. But at the same time, autologous stem cell transplantation is also faced with the age of patients, the influence of minimal residual disease (MRD) status before transplantation, chemotherapy dependence sensitivity, post-transplantation recurrence, post-transplantation granulosis infection and other problems.

In this study, we explored the efficacy and safety of autologous stem cell transplantation combined with Anti-CD19 CAR-T cells in the treatment of B-cell NHL in patients with B-NHL who achieved partial response (PR) in the interim assessment after 3-4 courses of first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their legal guardians voluntarily participate and sign the informed consent;
2. Male or female patients aged 18-70 years (including 18 and 70 years);
3. CD19+ B-NH was confirmed by pathology and histology, and the patient achieved a partial response (PR) by interim assessment after 3-4 courses of first-line chemotherapy;
4. B-cell non-Hodgkin lymphoma mainly includes the following two types:

(1) Diffuse large B-cell lymphoma (DLBCL); Mantle cell lymphoma (MCL); 5. Measurable or evaluable lesions; 6. The patient's main tissues and organs function well:

1. Liver function: ALT/AST < 3 times the upper limit of normal (ULN) and total bilirubin ≤34.2μmol/L;
2. Renal function: creatinine < 220μmol/L;
3. Lung function: indoor oxygen saturation ≥95%;
4. Cardiac function: left ventricular ejection fraction (LVEF) ≥40%. 7. The patient's peripheral shallow venous blood flow is smooth, which can meet the needs of intravenous infusion; 8. Patients with ECOG score ≤2 and expected survival time ≥3 months.

Exclusion Criteria:

1. Women who are pregnant (urine/blood pregnancy test positive) or breastfeeding;
2. Men or women who have planned to become pregnant within the last 1 year;
3. The patients were not guaranteed to take effective contraceptive measures (condoms or contraceptives, etc.) within 1 year after enrollment;
4. Patients had uncontrollable infectious diseases within 4 weeks prior to enrollment;
5. Active hepatitis B/C virus;
6. Hiv-infected patients;
7. Suffering from a serious autoimmune disease or immunodeficiency disease;
8. The patient is allergic to antibodies, cytokines and other macromolecular biological drugs;
9. The patient had participated in other clinical trials within 6 weeks prior to enrollment;
10. Systemic use of hormones within 4 weeks prior to enrollment (except for inhaled hormones);
11. Suffers from mental illness;
12. The patient has substance abuse/addiction;
13. According to the researchers' judgment, the patient had other conditions that were not suitable for inclusion.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | From 3 months to 1 year.
  Proportion of enrolled patients who achieved complete response after treatment

SECONDARY OUTCOMES:
overall survival | From 3 months to 1 year.
  The time interval between patient infusion of CAR-T and death from any cause or the end of follow-up.
Progression-free survival | From 3 months to 1 year.
  The time between treatment and observation of disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No